CLINICAL TRIAL: NCT03394950
Title: Butyphthalide in Combination With Recombinant Tissue Plasminogen Activator for Acute Ischemic Stroke (BRAIS)：a Pilot, Prospective, Random, and Double Blinded Multi-center Study
Brief Title: Butyphthalide in Combination With Recombinant Tissue Plasminogen Activator for Acute Ischemic Stroke
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hui-Sheng Chen (Other)
Responsible Party: Sponsor-Investigator, Hui-Sheng Chen, Professor, General Hospital of Shenyang Military Region
Organization: General Hospital of Shenyang Military Region (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: k201731
Record Dates: First submitted 2018-01-03; First posted 2018-01-09 (Actual); Last update posted 2021-06-02 (Actual); Status verified 2021-06

CONDITIONS: Stroke, Ischemic
Keywords: thrombolysis; Butyphthalide
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- rtPA combined with Butyphthalide (Experimental): Intravenous treatment with 25mg butyphthalide, followed by intravenous throbolysis with 0.9mg/kg rtPA. Next day, intravenous treatment with 25mg butyphthalide 2 times/day for 14 days, followed by oral butyphthalide capsule (0.2g 3 times/day) to 90 days after thrombolysis. Other treatments were done according to guidelines.
  Interventions: Drug: Butyphthalide combined with rtPA
- rtPA compared with placebo (Active Comparator): Intravenous treatment with placebo injection, followed by intravenous throbolysis with 0.9mg/kg rtPA. Next day, intravenous treatment with placebo injection 2 times/day for 14 days, followed by oral placebo capsule (3 times/day) to 90 days after thrombolysis. Other treatments were done according to guidelines.
  Interventions: Drug: rtPA

INTERVENTIONS:
Drug: Butyphthalide combined with rtPA — Intravenous treatment with 25mg butyphthalide, followed by intravenous throbolysis with 0.9mg/kg rtPA. Next day, intravenous treatment with 25mg butyphthalide 2 times/day for 14 days, followed by oral butyphthalide capsule (0.2g 3 times/day) to 90 days after thrombolysis. Other treatments were done according to guidelines.
  Arms: rtPA combined with Butyphthalide
Drug: rtPA — Intravenous thrombolysi with 0.9mg/kg rtPA, followed by other treatments according to guidelines
  Arms: rtPA compared with placebo

SUMMARY:
Acute ischemic stroke (AIS) is the most common type of stroke, which has high rate of morbidity, mortality and disability. A large number of studies have confirmed that the thrombolytic therapy can effectively open blood vessels and improve the functional prognosis of acute ischemic stroke. Therefore, all guidelines recommend giving thrombolysis treatment to acute ischemic stroke patients within 4.5 hours of onset. However, about 1/3 patients receiving thrombolysis will have good prognosis, while a large number of patients will still be disabled and even dead. How to improve the neurofunctional prognosis of thrombolytic patients has been a hot topic in the world.

Butyl phthalide is type I chemical drugs. Some multicenter randomized, double-blind, placebo-controlled clinical trials have showed that acute ischemic stroke patients taking butyl phthalide has better lateral branch circulation and living ability score than patients taking placebo. Besides, butyl phthalide treatment is safe. The animal experiment indicated that buphthalein could significantly improve secondary side branch circulation, recover the microarterial diameter of the soft meninges in the ischemic region and increase the blood flow rate.

Based on the discussion, we assume that: giving butyl phthalide to patients with acute ischemic stroke in advance, might promote and improve the formation of collateral circulation to freeze ischemia penumbra. Based on this hypothesis, we would like to explore the efficacy and safety of butyl phthalide combined with rtPA thrombolysis in the treatment of acute ischemic stroke.

ELIGIBILITY:
Inclusion Criteria:

1. Age >18 years;
2. Diagnosis of anterior circulation infarct;
3. First stroke onset or past stroke without obvious neurological deficit (mRS≤1);
4. Time from onset to treatment ≤4.5 hours;
5. SBP/DBP ≤ 180/110mmHg;
6. No hemorrhagic imaging changes showed in CT;
7. Signed informed consent by patient self or legally authorized representatives.

Exclusion Criteria:

1. History of stroke within 3 months;
2. History of intracranial hemorrhage;
3. Suspected subarachnoid hemorrhage;
4. Intracranial tumour, vascular malformation or arterial aneurysm;
5. Major surgery within 1 month;
6. Systolic pressure ≥180 mmHg or diastolic pressure ≥110 mmHg;
7. Platelet count < 100×109／L;
8. Heparin therapy or oral anticoagulation therapy within 48 hours;
9. Severe disease with a life expectancy of less than 3 months;
10. Blood glucose < 50 mg/dL (2.7mmol/L);
11. Patients who have received any other investigational drug or device within 3 months;
12. Researchers consider patients inappropriate to participate in the registry. -

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2018-05-25 (Actual); Primary Completion 2021-05-29 (Actual); Study Completion 2021-05-29 (Actual)

PRIMARY OUTCOMES:
Percentage of mRS score (0-2) (90 days) | 90 days
  Percentage of mRS score (0-2) at 90 days

CONTACTS AND LOCATIONS:
Overall Officials: chen huisheng, doctor, Study Director — General Hospital of Shenyang Military Region
Locations (1):
- General Hospital of ShenYang Military Region, Shenyang, China